CLINICAL TRIAL: NCT01042483
Title: Determination of Labor Progression Patterns Using Non-invasive, Ultrasound Based, Multiple Parameters+Continuous Vacuum Mode
Brief Title: Determination of Labor Progression Patterns Using Non-invasive, Ultrasound Based+Continuous Vacuum Mode
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Trig Medical Inc (Industry)
Responsible Party: Tzipi Yakoby, Director of Clinical Marketing, TrigMedical Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CLP003/2009
Record Dates: First submitted 2010-01-03; First posted 2010-01-05 (Estimated); Last update posted 2010-01-05 (Estimated); Status verified 2010-01

CONDITIONS: Pregnancy; Labor
Keywords: active stage; labor; progression; pregnant women during active phases of labor
MeSH Terms: conditions — Disease Progression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: LaborPro device — monitoring labor progression by using a new device The LaborPro system (Trig Medical Inc) allows determination of fetal head station and position using ultrasound and position tracking system.
  Other Names: LaborPro TrigMedical

SUMMARY:
The purpose of this study is to establish normograms of parameters measured by the LaborPro system, and to test the prediction of these parameters on labor progress and mode of delivery.

DETAILED DESCRIPTION:
Intrapartum assessment of the fetal head position and station, and cervical dilatation are essential for the management of labor. Precise knowledge of these parameters assists in the correct identification of normal versus abnormal labor progression patterns, and in case of the latter, indicates when medical or operative intervention may be required.

Digital examination remains the "gold standard" for evaluation of head station and position and cervical dilatation in pregnancy; however, it has inherent variability.

evaluations of the reliability of cervical dilatation assessment were performed initially in models, and more recently in patients during labor. Accuracy in models ranges from 51% to 59% and falls under 50% when evaluated in patients.

However, labor management has changed substantially since then. Induction of labor, oxytocin use, epidural analgesia, and fetal heart rate monitoring are very common in contemporary practice whereas breech vaginal delivery and mid forceps are rarely performed. The mean body mass of women is significantly higher than it was 50 years ago, which may contribute to the increased fetal size, and the second stage is prolonged, as it increasingly occurs with use of epidural analgesia. Some studies suggested that the Friedman curve was no longer appropriate for induced or actively managed labor.

In addition, once full dilatation is reached, although descent continues, monitoring of cervical dilation is no longer useful in the second stage. Descent in the second stage of labor is accompanied by rotation of the presenting part as it negotiates the pelvis. Friedman and Sachtleben showed that arrest of descent was frequently associated with fetal malpositions and suggested that abnormalities of rotation were important prognostic factors in the second stage.

The rates of caesarean section have been a major public health concern. Non progressive labor is the leading cause of primary C-sections in the US. It is well known that non-progressive labor is over diagnosed, and determination of the patterns of normal and abnormal labor is fundamental to the formulation of strategies to reduce caesarean section rates. In the US, the total cesarean delivery rate for 2005 rose to the highest level ever reported - 30.3%.After declining between 1989 and 1996, the cesarean rate has increased by 46 percent from the 1996 low of 20.7. The American College of Obstetricians and Gynecologists Task Force on Caesarian Delivery Rates (2000) recommended a C-section rate of 15.5% for nulliparous women for the US for the year 2010.

The LaborPro provides a tool for frequent non-invasive evaluation of head station and position, head descend, head descend during contraction, head position, and head rotation, without increasing the risk of maternal/fetal infection related to the number of vaginal examinations. In addition, a ruler-like determination of cervical dilatation is available during TVDE, as well as measurements of Pelvis diameters.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* Pregnant adult woman in labor
* Gestational age 37-42 wks
* Vertex presentation
* Willing to participate in the study and understands the study

Exclusion Criteria:

* Fetal malformations
* Fetal distress

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 450 (Estimated)
Dates: Start 2010-01; Primary Completion 2011-02 (Estimated); Study Completion 2011-02 (Estimated)

PRIMARY OUTCOMES:
Assessment of the LaborPro as a prediction tool of labor progression. by introducing extended labor curves. | 1 year

SECONDARY OUTCOMES:
Assessing the influence of obstetric and maternal parameters on the labor progression,relation between the pelvis diameters and Pubic Arch Angle measured by the LaborPro, and labor progression and mode of delivery,Maternal Satisfaction. | 1 year
Measurements of fetal head station and position during performing vacuum extraction delivery by attaching the positon sensor (1.3 mm) to the vacuum cup. | 1 year